CLINICAL TRIAL: NCT02033057
Title: Muscular Electrostimulation of the Sedated and Mechanically Ventilated Critically Ill Patient. Analysis of the Effect on Acquired Muscular Weakness and Its Clinical Consequences.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Paula Ramirez, doctor, Hospital Universitario La Fe
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pi12/01018
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2012-10

CONDITIONS: Polyneuropathy
Keywords: Muscular electrostimulation, mechanically ventilated, critically ill patients, muscular weakness.
MeSH Terms: conditions — Polyneuropathies; Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Muscular electrostimulation. (Experimental): The interventions is muscular electrostimulation.
  Interventions: Procedure: Muscular electrostimulation and percutaneus muscular biopsy.

INTERVENTIONS:
Procedure: Muscular electrostimulation and percutaneus muscular biopsy. — Muscular electrostimulation everyday and percutaneus muscular biopsy weekly.

SUMMARY:
Even 20-50% of patients under sedation and mechanical ventilation develops myopathy and / or neuropathy which difficulties both the process of extubation and the functional recovery. The objective of this project is to analyze the effect of muscle electrostimulation (ESM) on muscle weakness acquired in Intensive Care Unit (ICU) and its consequences. Study design: a single center, prospective, randomized trial to be held in the ICU of " Universitarian hospital La Fe" in collaboration with the service of Neurophysiology of the hospital. All patients undergoing sedation and mechanical ventilation (with an expected duration longer than 48h) and without any of the exclusion criteria detailed in the Methodology section will be included in the study. The intervention will consist of a muscular electrostimulation with the Super Pro Excel 70,UltratoneTM. The stimulation will be performed in 10 muscle groups (5 per side) following established protocols, at least 5 days a week. We will evaluate muscle strength by Medical Research Council scale, functional capacity by Barthel scale and Neurophaty Disability Scale, all clinical events will be collected and electrophysiologic, echographic and histologic parameters will be measured. The process of extubation will be performed following an established protocol, the duration will be collected as the same manner as ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Sedated and mechanically ventilated critically ill patients, more than 48 hours.

Exclusion Criteria:

* Body mass index > 45 or < 20 kg/m2.
* Pregnant.
* Epilepsia.
* Use muscular blocks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
muscular weakness | at the time of weaning, 30 days after extubation and one year after extubation.
  We measure the muscular weakness, with the medical research council scale.

SECONDARY OUTCOMES:
time of weaning | everyday

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario y Politécnico La Fe., Valencia, Valencia, Spain